CLINICAL TRIAL: NCT01742923
Title: Pharmacist Intervention Programme in Secondary Care to Improve Medication Adherence in Patients With Hypertension
Brief Title: Tailored Intervention to Improve Medication Adherence in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ulla Hedegaard, PhD student, MSc (pharm), Odense University Hospital, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AKF-384
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
Keywords: hypertension; medication adherence; motivational interviewing
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Placebo Comparator): Usual care
  Interventions: Behavioral: Usual care
- Complex tailored intervention (Experimental): The interventions consists of 3 elements:
  1. Medication review with recommendations focused on antihypertensives and statins and adherence to guidelines and patient´s adherence to medications
  2. Consultation with a pharmacist using motivational interviewing techniques
  3. Follow-up telephone calls one month and six months after inclusion
  Interventions: Behavioral: Complex tailored intervention

INTERVENTIONS:
Behavioral: Complex tailored intervention
  Arms: Complex tailored intervention
Behavioral: Usual care
  Arms: Usual care

SUMMARY:
Patients with hypertension have an increased risk of stroke and myocardial infarction. However, poor adherence to treatment with antihypertensives and lipid-lowering agents occurs frequently within this patient group. The purpose of this study is to investigate whether a complex tailored intervention in a hospital setting will lead to increased medication adherence and fewer cardiovascular events when compared to a usual care group. Interventions focus on motivational interviewing, medication review and telephone follow up.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 years or older

* Patients receiving ambulatory treatment for hypertension in a hospital setting
* The patient or a carer usually dispenses the patient's medications
* Patient lives in the Southern Region of Denmark
* Written consent

Exclusion Criteria:

* Lives in a care home or institution
* Receive dose dispensed medicine from a pharmacy
* Medicine is dispensed by a nurse in the patient's home
* Correctional mental health patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percent of patients that are at least 80% adherent (Medication possession rate > 0.8) to antihypertensives and statins | One year from inclusion

SECONDARY OUTCOMES:
Non-persistence with antihypertensives and statins measured by percent of patients that are not supplied with medications for more than three continuous months | One year from inclusion
Reduction in systolic and diastolic blood pressure | One year from inclusion
Composite endpoint (stroke, myocardial infarction or cardiovascular death) | One year from inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Result] Hedegaard U, Kjeldsen LJ, Pottegard A, Henriksen JE, Lambrechtsen J, Hangaard J, Hallas J. Improving Medication Adherence in Patients with Hypertension: A Randomized Trial. Am J Med. 2015 Dec;128(12):1351-61. doi: 10.1016/j.amjmed.2015.08.011. Epub 2015 Aug 21. PMID 26302142
- [Result] Hedegaard U, Hallas J, Ravn-Nielsen LV, Kjeldsen LJ. Process- and patient-reported outcomes of a multifaceted medication adherence intervention for hypertensive patients in secondary care. Res Social Adm Pharm. 2016 Mar-Apr;12(2):302-18. doi: 10.1016/j.sapharm.2015.05.006. Epub 2015 May 18. PMID 26088274